CLINICAL TRIAL: NCT04171063
Title: Safety and Efficacy of a Modular and Adjustable Chest Compressor Model for Conservative Treatment of Pectus Carinatum: a Multicenter Study
Brief Title: Chest Compressor for Conservative Treatment of Pectus Carinatum: a Multicenter Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Miguel L. Tedde, Staff Physician, General Thoracic Surgery Department, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USaoPauloGH
Record Dates: First submitted 2019-11-07; First posted 2019-11-20 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Pectus Carinatum, Chondromanubrial
Keywords: Braces; Conservative treatment; Thoracic wall; Pectus carinatum
MeSH Terms: conditions — Pectus Carinatum

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to use the thoracic compressor for 16 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bracing arm (Other): Patients that will be using the thoracic compressor
  Interventions: Device: Thoracic compressor

INTERVENTIONS:
Device: Thoracic compressor — The intervention is the use of the thoracic compressor for the conservative treatment of pectus carinatum

SUMMARY:
Pectus carinatum (PC) is a congenital deformity of the chest wall whose prevalence is 0.6% of the population and although it does not cause cardio respiratory physiological damage, it has profound psychological effects on young people. Its treatment today is still primarily surgical in our country, despite the fact that conservative treatment by chest compression may be effective in the chondrogladiolar variant, which represents 90% of cases of PC. The aim of the present study is to conservatively treat a series of 60 patients using a new modular and adjustable chest compressor model to assess the effectiveness of this chest compressor in the noninvasive treatment of PC; and also assess the safety of such treatment by the rate of adverse events occurring during treatment. Secondary objectives will be to evaluate the adherence that PC patients have to this type of treatment by quantifying the number of hours of use per day, besides evaluating the chest compressor and its components for durability and resistance as a device for continuous use.

ELIGIBILITY:
Inclusion Criteria:

* Pectus carinatum condrogladiolar Variant
* No other comorbidities that could interfere with the use of compressor

Exclusion Criteria:

* Marfan Syndrome
* Active cardiovascular disease
* Significant scoliosis or thoracic deformity
* Important obesity
* Pectus carinatum chondromanubrial variant
* Poor commitment to protocol by both research participant and parents

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment efficiency in repairing the pectus carinatum | 16 months
  The anthroprometric measures in centimeters of the thoracic cage will be taken before and after the treatment to evaluate the effectiveness of the chest compressor in repairing the pectus carinatum
Treatment safety | 16 months
  The adverse events that can possibly occur during treatment will be recorded in the patients using the chest compressor for pectus carinatum repair

SECONDARY OUTCOMES:
Treatment adherence | 16 months
  The number of hours of daily use of the chest compressor will be recorded as a measurement of the level of adherence to the chest compressor treatment
Device durability | 16 months
  The mechanic problems presented by the chest compressor as fractures, screw loosening or fastener break will be recorded as a durability and strength measure of the chest compressor and its components.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Tedde, MD, PhD, Principal Investigator — Instituto do Coracao (InCor) HCFMUSP
Locations (4):
- Brazil (4):
  - Hospital de Clinicas da Faculdade de Botucatu, Botucatu, São Paulo
  - Hospital das Clinicas da Unicamp, Campinas, São Paulo
  - Instituto do Coracao (InCor) HCFMUSP, São Paulo, São Paulo
  - Hospital das Clinicas da USP Ribeirao, Ribeirão Preto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kelly RE Jr, Lawson ML, Paidas CN, Hruban RH. Pectus excavatum in a 112-year autopsy series: anatomic findings and the effect on survival. J Pediatr Surg. 2005 Aug;40(8):1275-8. doi: 10.1016/j.jpedsurg.2005.05.010. PMID 16080931
- [Result] Shamberger RC. Congenital chest wall deformities. Curr Probl Surg. 1996 Jun;33(6):469-542. doi: 10.1016/s0011-3840(96)80005-0. No abstract available. PMID 8641129
- [Result] Kelly RE Jr, Shamberger RC, Mellins RB, Mitchell KK, Lawson ML, Oldham K, Azizkhan RG, Hebra AV, Nuss D, Goretsky MJ, Sharp RJ, Holcomb GW 3rd, Shim WK, Megison SM, Moss RL, Fecteau AH, Colombani PM, Bagley TC, Moskowitz AB. Prospective multicenter study of surgical correction of pectus excavatum: design, perioperative complications, pain, and baseline pulmonary function facilitated by internet-based data collection. J Am Coll Surg. 2007 Aug;205(2):205-16. doi: 10.1016/j.jamcollsurg.2007.03.027. Epub 2007 Jun 21. PMID 17660066
- [Result] Desmarais TJ, Keller MS. Pectus carinatum. Curr Opin Pediatr. 2013 Jun;25(3):375-81. doi: 10.1097/MOP.0b013e3283604088. PMID 23657247